CLINICAL TRIAL: NCT04546269
Title: Fully Guided Versus Conventionally Guided Implant Placement by Dental Students. A Randomized Controlled Trial
Brief Title: Fully Guided Versus Conventionally Guided Implant Placement by Dental Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Simon Storgård Jensen, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19037743
Record Dates: First submitted 2020-08-28; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Implant Dentistry; Guided Implant Placement; Single tooth implant; Computer-guided surgery
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: The assesor was blinded to the group allocation of the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fully-guided (Experimental): Single-tooth implant placed using a fully computer-guided approach
  Interventions: Procedure: Fully-guided vs. conventionally guided implant placement
- Conventionally guided (Active Comparator): Single-tooth implant placed using a conventionally guided approach
  Interventions: Procedure: Fully-guided vs. conventionally guided implant placement

INTERVENTIONS:
Procedure: Fully-guided vs. conventionally guided implant placement — Patients randomized to implant placement planned virtually based on a CBCT and a surface scan vs. implant placement based on a wax-up on gypsum casts

SUMMARY:
Patients where placement of a single implant will be treated by senior dental students under close supervision of experienced spcialists. All implant treeatments will be categorized as "straight forward"according to the SAC classification. The patients will be randomized to have the implants placed using a fully guided or a convetionally guided protocol.

Outcome parameters include accuracy of implant placement compared to an ideal implant position, patient- and student-reported outcome.

DETAILED DESCRIPTION:
Study design and participants The study is designed with two commonly used procedures for implant placement. Two well-known, but different workflows are used: a digital using primarily a digital workflow and a conventional workflow using primarily an analog procedure. In our daily student education, the latter has been used, but to examine the feasibility and quality of using a full digital work, the present study will compared two accepted and documented workflows. For making a reliable comparison, a prospective, randomized clinical study is planned within our normal schedule for student education. Thirty-six patients are already recruited and pre-screened to clinical teaching in implant dentistry on from the September to December 2019 on Department of Odontology. All 36 patients in the need of implant-supported single tooth restorations and without any contraindications for implant dentistry. All cases are selected to be "straight-forward" cases possible to be rehabilitated by dental students.

Sample calculation (Power of the study): A sample size of 28 subjects (14 in each group) is needed to detect a difference in patient-reported outcome (VAS-scale values for digital versus analog impression) of 30 % , with a 5 % risk of type I and 20 % risk of type II errors and SD = 2. With a maximum drop-out of up to 8 patient a sample size of 36 is endeavored.

The inclusion criteria for this study are the following:

* Patients of more than 18 years of age
* Patients with a need of one or more single-tooth implants in the molar or the premolar region
* Natural healthy neighboring teeth without need of restorations
* Sufficient bone-volume for placing an implant without bone- or soft tissue augmentation

Exclusion criteria are the following:

* Heavy smokers (more than 10 cigarettes per day)
* Uncontrolled diabetes
* Metabolic bone disorders
* History of radiotherapy of the head and neck
* Recent chemotherapy
* Use of drugs inﬂuencing bone or soft tissue healing (e.g. high doses of antiresorptive medication, steroids or anti-inflammatory drugs)
* Additional oral surgery in the region of interest

Intervention The patients in the digital group (test) will be treated following a digital workflow and the analog group (control) will be treated with the same workflow as the students have used the last three years in the student educational program.

Workflow Study groups Digital Test (T) , n=18 Analog Control (C), , n=18 Pre-examination CBCT, Limited to two neighboring teeth at both side or 4 teeth mesially for the distal implants.

A bite index with a thickness of 3-5 mm will be used to stabilize and separate the jaws during scanning.

IOS (Digital impression) CBCT, Limited to two neighboring teeth at both side or 4 teeth mesially for the distal implants.

A bite index with a thickness of 3-5 mm will be used to stabilize and separate the jaws during scanning.

Conventional analog impression Planning The SIMPLANT™ (Dentsply) software will be used. The DCOM-file from CBCT and STL-file from IOS will be downloaded to Dentsply, Simplant Academy service center. In cooperation with dentists and students, the most optimal placement of implants will be planned. Based on this treatment plan, a "Tooth-supported Simplant Guide" for surgical procedure will be milled. The stone model prepared from the conventional analog impressions will be used. In the toothless regions, an acrylic tooth of the proper size will be placed on the most optimal position and fixed on the stone model with wax-up technique.

A customized acrylic surgical guide will be ordered and produced by dental technician. The CBCT will be used for planning the best position of implants and will be used for visual guidance during implant insertion (Soft ware: Planmeca Romexis®).

Implant insertion

Computer-guided implant surgery The tooth-supported surgical guide with metallic sleeves covering the occlusal plane of four teeth in the same jaw region will be used. Analog surgical guide The tooth-supported surgical guide without metallic sleeves covering the occlusal plane of four teeth in the same jaw region will be used.

Implants Astra Tech Osseospeed EV ® , non-submerged Astra Tech Osseospeed EV®, non-submerged Impression for prosthetic part IOS and conventional impression; IOS:for prosthetic construction. The other impression technique: for comparison of patient experience between the two methods. IOS and conventional impression Conventional impression: for prosthetic construction. The other impression technique: for comparison of patient experience between the two methods.

Color selection of crowns IOS of buccal aspect of neighboring teeth Color scale: Lumin Vacuum, Vitapan Fabrication of screw-retained crown-abutments CAD/CAM, stereolithograpic model based on IOS Abutment: Atlantis® Crown abutment (Titanium) using porcelain fused to metal CAD/CAM, gypsum cast models, based on conventional impression Abutment: Atlantis® Crown abutment (Titanium) using porcelain fused to metal CBCT: Cone Beam Computed Tomography OP: Orthopantomogram IOS: Intraoral scanning CAD/CAM: Computer-Aided Design/ Computer-Aided Manufacturing

Randomization Thirty-six sealed, opaque envelopes containing the letters T or C, representing test (fully digital workflow) and control (conventional workflow) group, will be used. At the first visitation at the Section of Oral Rehabilitation, patients will be informed about the allocation and the treatment procedure. The patients will draw an envelope and the name of the participants will be written on the envelope and the envelope will be opened. Clinical photographs of smile line, front region, premolar/molar region at both sides and occlusal planes will be taken.

Surgical procedures After a primary visitation of the patients by an oral surgeon at the Section of Oral Surgery. In both test (nT=18) and control group (nC=18) Cone Beam Computed Tomography (CBCT; Viso Planmeca, Finland) will be taken of the implant region and the SIMPLANT™ (Dentsply) software will be used to plan the implant position. In the test group a fully guided procedure with a surgical guided with metal sleeves produced based on the STL file from the software. In the control group, an analog surgical guide without metallic sleeves and with relatively high freedom of movements will be used be the student during implant surgery. The patients group C and T will be going through implant insertion procedures as listed in Table 1. The surgical guides produced for the group T and C will be used during the surgical procedure of implant insertion. After healing of implants, the patients will be referred to the Section of Oral Rehabilitation for prosthetic treatment.

Prosthetic procedures Ten to fourteen weeks after implant placement, the implants will be clinically tested for osseointegration, and impressions will be taken. To evaluate the patient satisfaction and convenience with the digital versus the analog technique, all 36 patients will try the digital as well as the analog impression. CEREC intraoral scanners will be used for the digital technique, and conventional impression techniques will be used for the analog technique. For intraoral scanning, scan bodies will be used, and the implant region, antagonistic teeth and occlusal registrations will be performed. The analog impressions include the use of implant pick-ups and Impregum (3M, ESPE) for impression of the actual arch, Blue Mousse (Parkell, USA) for occlusal registration, and Alginate (ALGINoplast®, Kulzer GmbH, Hanau, Germany) for the opposite arch.

The prosthetic restorations will be screw-retained crown-abutments designed using CAD/CAM technique on either stereolithographic models for the test participants (digital technique), or on gypsum cast-models for the participants in the control group (conventional technique) . The participants will be recalled to follow-up examinations 4 weeks after crown fixation.

Outcome - Evaluation

1. Accuracy of guided implant surgery After implant placement all 36 patients will have a new CBCT of the implant region and an overlay of the two CBCT´s (before and after implant placement) will be used for measuring deviations between the planned implant position and the real implant position: Apical deviation (mesio-distally, bucco-lingually), Marginal deviation (mesio-distally, bucco-lingually) to test for accuracy of the two methods. Measurements will be performed in the computer software, where DICOM files from CBCT´s can be transferred to STL-files from IOS's.
2. Prosthetic quality of the implant-supported restoration

   Technical outcome: The following prosthetic quality criteria is registered for the crown-abutments screw into the fixtures:
   * Occlusion points

     * infra-occlusion: no occlusal point on a 40 µm thick foil
     * supra-occlusion: to hard occlusal points evaluated with a 40 µm thick foil
   * Contact points (evaluated with a dental floss)

     * Mesial contact (hard, light or no interproximal contact)
     * Distal contact (hard, light or no interproximal contact)
3. Aesthetic outcome Will evaluated with the Copenhagen Index score, including score for harmony/symmetry, crown color, crown morphology, mucosal discoloration and papillas (Dueled, Gotfredsen, Damsgaard, & Hede, 2009; Hosseini & Gotfredsen, 2012)
4. Patient satisfaction and convenience of the two procedures. Qualitative and quantitative evaluation of the two procedures.
5. Process evaluation i) Observation (quality description) of the surgical procedures (time used and challenges with the two procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 18 years of age
* Patients with a need of one or more single-tooth implants in the molar or the premolar region
* Natural healthy neighboring teeth without need of restorations
* Sufficient bone-volume for placing an implant without bone- or soft tissue augmentation

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes per day)
* Uncontrolled diabetes
* Metabolic bone disorders
* History of radiotherapy of the head and neck
* Recent chemotherapy
* Use of drugs inﬂuencing bone or soft tissue healing (e.g. high doses of antiresorptive medication, steroids or anti-inflammatory drugs)
* Additional oral surgery in the region of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Linear and angular accuracy of implant placement | 1 year
  Linear (in mm) and angular (in degrees) deviations from an ideal implant position determined by three experienced investigators.

SECONDARY OUTCOMES:
Patient-reported outcome | 1 year
  OHIP questionnaire filled in by the patients with four ratings of 14 questions: Seldom, Sometimes, Often, Always

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, School of Dental Medicine, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No